CLINICAL TRIAL: NCT03596502
Title: Safety and Effectiveness of Direct Oral Anticoagulants for Stroke Prevention in Non-valvular Atrial Fibrillation: a Multi-database Cohort Study with Meta-analysis (DOACs Vs Warfarin)
Brief Title: Direct Oral Anticoagulants in Patients with Atrial Fibrillation (DOACs Vs Warfarin)
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q16-13B
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation; Ischemic Stroke; Systemic Embolization; Major Bleed; Myocardial Infarction; All-cause Mortality
Keywords: Direct oral anticoagulants; Safety; Atrial fibrillation; Ischemic stroke; Systemic embolization
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Myocardial Infarction | interventions — N(4)-oleylcytosine arabinoside; apixaban; Dabigatran; Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Direct oral anticoagulants (DOACs): Patients diagnosed with non-valvular atrial fibrillation who initiated their oral anticoagulation with a DOAC (apixaban, dabigatran or rivaroxaban) at cohort entry date, and did not have a previous prescription for any oral anticoagulant in the prior year.
  Interventions: Drug: Direct oral anticoagulants (DOACs)
- Warfarin: Patients diagnosed with non-valvular atrial fibrillation who initiated their oral anticoagulation with warfarin at cohort entry date, and did not have a previous prescription for any oral anticoagulant in the prior year.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Direct oral anticoagulants (DOACs) — Exposure to DOACs will be defined as a new prescription for apixaban (ATC B01AF02), dabigatran (ATC B01AE07), or rivaroxaban (ATC B01AF01) at cohort entry date in patients diagnosed with non-valvular atrial fibrillation.
  Other Names: Eliquis, Pradaxa, Xarelto
  Groups: Direct oral anticoagulants (DOACs)
Drug: Warfarin — Exposure to warfarin will be defined as a new prescription for warfarin (ATC B01AA03) at cohort entry date in patients diagnosed with non-valvular atrial fibrillation.
  Other Names: Coumadin
  Groups: Warfarin

SUMMARY:
The purpose of this study is to assess safety and effectiveness of direct oral anticoagulants (DOACs) and warfarin for stroke prevention in patients with non-valvular atrial fibrillation (AF). The comparison of DOACs versus oral vitamin K antagonists, in particular warfarin, is of interest.

The investigators will carry out separate population-based, matched cohort studies, using health administrative databases in seven Canadian provinces. New users of oral anticoagulants (DOACs or warfarin) for stroke prevention in non-valvular AF will be eligible to enter the cohorts. Follow-up will continue until a hospitalization or emergency department visit for a stroke. The results from the separate sites will be combined by meta-analysis to provide an overall assessment of the safety and effectiveness of the different anticoagulation regimens in stroke prevention in AF.

The investigators hypothesize that DOACs and warfarin will have similar safety and effectiveness profiles.

DETAILED DESCRIPTION:
The objective of this study is to assess safety and effectiveness of direct oral anticoagulants (DOACs) and warfarin for stroke prevention in patients with non-valvular atrial fibrillation (AF).

A common-protocol approach will be used to conduct retrospective cohort studies using administrative health care data from seven Canadian provinces (Alberta, British Columbia, Manitoba, Nova Scotia, Ontario, Quebec, Saskatchewan). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. The data in Alberta, Nova Scotia, and Ontario will be restricted to patients aged 65 years and older, as prescription data are not available for younger patients.

In each jurisdiction, the investigators will assemble a base cohort that includes all patients newly prescribed an oral anticoagulant (DOAC or warfarin) for stroke prevention in AF. Study period will be from the date of the first DOAC approval for stroke prevention in AF at each site to the date of latest data availability at each site. All patients newly dispensed an oral anticoagulant (i.e. with no prescription for any oral anticoagulant in the prior year) with a diagnosis of AF within the 3 years prior to the date of the prescription will be eligible to be included into the study cohorts, given they present no exclusion criteria. The date of study cohort entry will be defined by the dispensation date of the newly prescribed oral anticoagulant. Patients will be censored at the earliest of death, end of healthcare coverage, switch from DOAC to warfarin, switch from warfarin to DOAC, initiation of hemodialysis or heart valve surgery, or the end of the study period, whichever occurs first.

Exposure to a DOAC will be defined as a new prescription for a DOAC (apixaban, dabigatran, rivaroxaban) on the date of cohort entry. Exposure to warfarin will be defined as a new prescription for warfarin on the date of cohort entry. The investigators will use an analysis analogous to an intention-to-treat approach. The primary outcome will be defined as a hospitalization or emergency department visit for ischemic stroke or systemic embolization. The secondary outcomes will be: 1) major bleeding; 2) a composite of stroke (ischemic or hemorrhagic), systemic embolization, major bleeding or all-cause mortality; 3) myocardial infarction; 4) gastrointestinal bleeding; 5) intracranial bleeding; and 6) all-cause mortality.

The study cohort will be analyzed using a matched cohort design, where DOAC users will be matched 1:1 to warfarin users on sex, age, cohort entry date, and propensity score (which will be constructed using a multivariable logistic regression model estimating the odds of being treated with DOACs, while adjusting for a number of pre-identified covariates to account for baseline differences at the time of cohort entry). Cox-proportional hazards regression models will be used to estimate adjusted hazards ratios (HRs) and corresponding 95% confidence intervals (CIs) for ischemic stroke or systemic embolization in the three cohorts. Meta-analyses of the site-specific results will be performed using random effects models. As secondary analyses, the composite outcome will be stratified by age (<85 and ≥85) and sex. In addition, an as treated analysis using inverse probability of censoring weights (IPCW) will be performed to account for non-random censoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new prescription for an oral anticoagulant that had a diagnosis of atrial fibrillation or atrial flutter within the 3 years prior to the date of the prescription
* Patients aged 18 years or older (except Alberta, Nova Scotia, and Ontario, where patients will be aged at least 66 years or older)

Exclusion Criteria:

* Patients with less than one year of data availability prior to cohort entry
* Patients with a diagnosis of valvular disease (including rheumatic heart disease) or prior cardiac valve surgery
* Patients with a diagnosis of venous thromboembolic disease in the year prior to cohort entry
* Patients who underwent hemodialysis in the 90 days prior to cohort entry
* Patients with a hip, femur, or knee surgery in the 30 days prior to cohort entry
* Patients with a diagnosis of antiphospholipid syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a study cohort that includes all patients newly anticoagulated from the date of the first DOAC approval for stroke prevention in AF (in each site) to the date of the latest data availability at each site, that had a diagnosis of AF within the 3 years prior to the date of the prescription.
Sampling Method: Probability Sample
Enrollment: 402764 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke (IS) or systemic embolization (SE) | Patients will be followed from date of first DOAC or warfarin prescription (cohort entry date) until a hospitalization or ED visit for IS or SE, censoring due to death, end of healthcare coverage, or for up to 65 months, whichever occurs first.
  Patients hospitalized or visiting the emergency department (ED) for a stroke or a systemic embolization recorded as the most responsible diagnosis in either the discharge abstract or hospitalization record with the following ICD codes:
  Ischemic stroke:
  ICD-9 codes: 434.x; ICD-10 codes: I63.x, I64.x
  Systemic embolization:
  ICD-9 codes: 444.x; ICD-10 codes: I74.x

SECONDARY OUTCOMES:
Major bleeding | Patients will be followed from date of first DOAC or warfarin prescription (cohort entry date) until a hospitalization or ED visit for major bleed, censoring due to death, end of healthcare coverage, or for up to 65 months, whichever occurs first.
  Patients hospitalized or visiting the emergency department (ED) for a major bleed composite recorded as the most responsible diagnosis in either the discharge abstract or hospitalization record with the following ICD codes:
  Intracranial bleeding (including hemorrhagic stroke):
  ICD-9 codes: 430.x, 431.x, 432.x; ICD-10 codes: I60.x, I61.x, I62.x
  Gastrointestinal bleeding:
  ICD-9 codes: 456.0, 531.0, 531.2, 531.4, 531.6, 532.0, 532.2, 532.4, 532.6, 533.0, 533.2, 533.4, 533.6, 534.0, 534.2, 534.4, 534.6, 569.3, 578.x; ICD-10 codes: I85.0, I98.3, K25.0, K25.2, K25.4, K25.6, K26.0, K26.2, K26.4, K26.6, K27.0, K27.2, K27.4, K27.6, K28.0, K28.2, K28.4, K28.6, K29.0, K55.21, K62.5, K63.81, K92.0, K92.1, K92.2
  Ocular bleeding:
  ICD-9 codes: 362.81, 363.6x, 376.32, 379.23, 377.42; ICD-10 codes: H31.3, H35.6, H43.1, H45.0
  Other bleeding causing ED visit or hospitalization:
  ICD-9 codes: 459.0, 596.7, 599.7, 627.1, 719.1, 729.92, 784.7, 784.8, 786.3; ICD-10 codes: D68.3, K66.1, M25.0x, N02.x
All-cause mortality | Patients will be followed from date of first DOAC or warfarin prescription (cohort entry date) until death, end of healthcare coverage, or for up to 65 months, whichever occurs first.
Myocardial infarction | Patients will be followed from date of first DOAC or warfarin prescription (cohort entry date) until a hospitalization for a myocardial infarction, censoring due to death, end of healthcare coverage, or for up to 65 months, whichever occurs first.
  Patients hospitalized for a myocardial infarction recorded as the most responsible diagnosis in hospitalization record with the following ICD codes:
  ICD-9 codes: 410.x; ICD-10 codes: I21.x

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Durand, MD, MSc, FRCPC, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre de recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durand M, Schnitzer ME, Pang M, Carney G, Eltonsy S, Filion KB, Fisher A, Jun M, Kuo IF, Renoux C, Paterson JM, Quail J, Matteau A; Canadian Network for Observational Drug Effect Studies Investigators. Comparative effectiveness and safety of direct oral anticoagulants versus vitamin K antagonists in nonvalvular atrial fibrillation: a Canadian multicentre observational cohort study. CMAJ Open. 2020 Dec 18;8(4):E877-E886. doi: 10.9778/cmajo.20200055. Print 2020 Oct-Dec. PMID 33355273
- See also: This is the website describing the general functions of the organization, other CNODES projects, and investigator profiles. — http://www.cnodes.ca